CLINICAL TRIAL: NCT05566782
Title: Cross-sectoral Rehabilitation After Stroke (CRES)
Acronym: CRES
Status: Active, not recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Tafdrup Notkin, Principal Investigator, Nordsjaellands Hospital
Other Study IDs: CRES&SENS
Record Dates: First submitted 2022-09-26; First posted 2022-10-04 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Neurological Rehabilitation; Patient Involvement
MeSH Terms: conditions — Stroke; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CRES-participants: The participants in this cohort will start rehabilitation during their inhospital stay and continue the rehabilitation course during discharge to municipality.
  The rehabilitation will consist of physical exercise and measurements in relation to accelerometry, physical function and qualitative interviews regarding goal for rehabilitation.

SUMMARY:
Prospective cohort study during post stroke rehabilitation in hospital and municipality. Participants will be measured with accelerometers, tests in relation to physical function and qualitative interviews.

DETAILED DESCRIPTION:
During and after hospitalization, patients with stroke are subjected to early rehabilitation starting at the hospital stay and continuing after discharge to a municipality. However, the continuity and adherence across sectors is challenged by different locations for the rehabilitation and time gaps from discharge to start in municipality.

This project focuses on the physical activity of patients with stroke measured with 3D accelerometry, the physical performance of the patients measured using the 30 second Chair Stand Test, balance measured with Bergs Balance Scale and health-related quality of life (HRQoL) measured with the 5-level version of European Quality of Life (EQ5D-5L). Furthermore, the patient perspectives and experiences with the rehabilitation plans are explored in semi-structured interviews at the end of the project.

The municipalities in Nordsjælland have been informed regarding the project and all their approvals have been collected prior to expected start in fall 2022. The heads of rehabilitation in the municipalities have approved participation in the research project with regards to follow-up of patients. The municipalities will support the data collection process with a therapist from each municipality working with quality control of the rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age;
* Hospitalized at Nordsjællands Hospital (NOH) with acute stroke;
* Discharged from the Department of Neurology NOH with a general rehabilitation plan to one of the eight surrounding municipalities (Hillerød, Allerød, Gribskov, Helsingør, Hørsholm, Halsnæs, Frederikssund Fredensborg);
* able to give written informed consent;

Exclusion Criteria:

* Poor Danish language skill;
* Patients refusing any rehabilitation or medically assessed as inevitably dying within 12 weeks;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity is based on medical records and personal identification number
Study Population: Participants will be recruited by the PhD-student Gabriel Tafdrup Notkin (GTN) in collaboration with the Department of Neurology. Potential participants will be approached during admission at the Department of Neurology, NOH.
  Potential participants will be informed about the study orally and in writing. Patients will be informed that participation is voluntary and that they can withdraw from the study at any time. There will be an opportunity for reflection time and for the patient to discuss the decision to participate with relatives or caregivers. If the patient wishes to participate in the study, written consent will be obtained in the form of a completed consent form from the patient and relatives.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2025-10-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity measured by step counts and intensity minutes during the day (raw acceleration per time cycle) | 10-14 days from hospital discharge til start of rehabilitation in municipality
  3D Accelerometers able to capture the daily physical activity performed by the participants in terms of intensity minutes and daily step counts (physiological parameter)
Change in physical function (30 second chair stand test) | At four timepoints during rehabilitation. Anticipated days for testing: day 1, day 4, day 11, day 95
  Tests performed during in hospital stay and at discharge and at start/end of rehabilitation
Change in balance (Bergs Balance Scale) | At four timepoints during rehabilitation. Anticipated days for testing: day 1, day 4, day 11, day 95
  Tests performed during in hospital stay and at discharge and at start/end of rehabilitation in municipality. Scores registered in ordinal scale from 0-56 with higher scores indicating lower risk of fall. Bergs Balance Scale consists of 14 test items each with scores ranging from 0, 1, 2, 3 and 4.
Change in Health Related Quality of Life (EQ5D-5L) | Measurement at the start of rehabilitation (day 1) and at the anticipated end of rehabilitation (day 95)
  Measurements with EQ5D-5L send electronically to participants with REDcap system

SECONDARY OUTCOMES:
Severity of stroke (Scandinavian Stroke Scale) | within 24 hours of admission
  Registration from participants medical records. Scores reported in ordinal scale from 0-58 with higher scores indicating less severe impairment form stroke.
  Overall categories; mild: 43-58 moderate: 26-42 severe: 0-25
Rate of dependence post stroke evaluated by modified Rankin Scale (mRS) | Measurement at the discharge from hospital stay (anticipated day 4)
  Evaluation performed by primary investigator with participant. Scores in ordinal scale ranging from 0-6 with higher scores indicating worse outcomes post stroke.
Demographic variables | Measurement at the start of rehabilitation (anticipated day 1 of hospital admission)
  age, gender, body mass index, marital status, level of education, employment

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel T Notkin, MSc.PT., Principal Investigator — Physiotherapist, Department of Neurology
Locations (1):
- Nordsjællands Hospital Department of Neurology, Hillerød, Denmark